CLINICAL TRIAL: NCT00438854
Title: Phase II Study of Dasatinib (BMS-354825) in Relapsed Chronic Lymphocytic Leukemia
Brief Title: Dasatinib in Relapsed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Philip C. Amrein, M.D., Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-211; CA 180-045
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: dasatinib; BMS-354825; CLL; SLL; LYN kinase
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Dasatinib

ARMS (1):
- Dasatinib treatment (Experimental): All patients were treated with dasatinib pills by mouth as treatment.
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Taken orally once daily. Participants may continue on study treatment as long as there is no disease progression or serious side effects.

SUMMARY:
The purpose of this research study is to see if Dasatinib is effective and safe to give to people with relapsed chronic lymphocytic leukemia (CLL) and to determine the effects of the drug on LYN kinase activity in blood and bone marrow. Recent research shows that a key enzyme in CLL cells is responsible for cell survival. This enzyme is called LYN kinase. Laboratory studies show that inhibition of LYN kinase in CLL cells results in the death to CLL cells. Dasatinib has the ability to inhibit LYN kinase and, therefore, should have some effect on CLL cells.

DETAILED DESCRIPTION:
* After the screening procedures confirm that the participant is eligible and willing to participate in the research study, they will have the following tests and procedures.
* Dasatinib is given orally once daily. Each participant will have a pill diary to record doses and any missed doses. All necessary drug refills will be given during clinic appointments, at which time the pill diary and any unused study drug will be returned.
* During the first month of study treatment the participant will come to the clinic at the following intervals: Day 1: An EKG will be performed two hours after the first dose of medication; Days 3-8: Blood samples will be drawn once between days 3-8; Weeks 2-4: A physical examination, EKG and blood samples will be drawn once a week.
* Beginning with the second month of study treatment, participants will come to the clinic monthly for up to two years. The following tests and procedures will be done; physical examination (monthly), blood work (monthly), pregnancy test (monthly), EKG (monthly for 6 months, then when medically indicated), CT of the neck, chest and abdomen (every 2 months for 6 months, then once every 6 months), at the end of month 2, additional blood will be drawn for research testing.
* Participants can continue to take the study drug for up to two years as long as their disease does not progress and they are not experiencing any serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* CLL/SLL with cells positive by flow cytometry (or immunostaining) for CD19, CD23 and CD. Patients may be CD23 negative as long as they are also cyclin D1 negative.
* Must have failed at least 1 prior fludarabine containing regimen or have failed at least 2 non-fludarabine containing regimens or have a contraindication to fludarabine use
* ECOG performance status of 2 or better
* Adequate organ function to tolerate chemotherapy
* Adequate method of contraception

Exclusion Criteria:

* Pregnant or breast-feeding women
* Uncontrolled angina within 3 months
* Diagnosed or suspected congenital long QT syndrome
* History of clinically significant ventricular arrhythmias
* Prolonged QTc interval on pre-entry electrocardiogram
* Uncontrolled hypertension
* Drugs that are generally accepted to have a risk of causing Torsades de Pointes
* Patient known to be HIV positive
* Known significant bleeding disorder unrelated to CLL
* Drugs that interfere with platelet function or coagulation must be stopped at least 7 days prior to entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-12; Primary Completion 2010-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Amrein, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Started recruitment 12/2006 and ended recruitment 12/2008. Patients were recruited from the clinics of the Massachusetts General Hospital and the Dana Farber Cancer Institute.
Pre-assignment Details: Patients signing the consent form were screened for eligibility. If eligible, they were started on protocol. This is a single-arm protocol.
Period: Overall Study
Arm/Group | Dasatinib Treatment
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Overall objective response rate in terms of complete response, nodular partial response, and partial response to treatment. Objective response is when a biopsy shows. In general response is defined as the following (not complete criteria):
  Complete response (CR) requires all of the following for a period of at least 2 months:
  * Absence of lymphadenopathy
  * No hepatomegaly or splenomegaly
  * Absence of constitutional symptoms
  * Normal complete blood count
  Nodular partial response (nPR): Met the criteria for CR, but had residual bone marrow biopsy nodules as the only evidence of disease
  Partial response (PR): requires at least the following:
  * 50% decrease in peripheral blood lymphocyte count
  * 50% reduction in lymphadenopathy
  * 50% reduction in the size of the liver and/or spleen
Time Frame: 2 years
Measure: Number; unit: participants who responded
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 15
participants who responded | 3
Statistical Analysis 1: Comparison: Dasatinib Treatment; The primary measures of efficacy of tumor response were: complete remission (CR), nodular partial remission (nPR), or partial remission (PR), as per NCI-WG criteria. The true ORR is reported as percentage and 90% CI calculated using the binomial exact test. Time to treatment failure (TTF) was defined from the date on study to date of progression, death in remission, initiation of non-protocol therapy in the absence of progression, or censored on the last visit; Test type: Superiority or Other; Estimating proportion of responders = 0.20

2. Secondary Outcome: Complete Response Rate
Description: The number of participants with a 100% reduction in nodal mass.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 15
Participants | 0

3. Secondary Outcome: Median Time to Disease Progression
Description: The median time to disease progression, measured from the start of treatment.
Time Frame: 1 year
Measure: Median (Full Range); unit: Months
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 15
Months | 7.5 [0.6 to 34.4]

4. Secondary Outcome: Median Overall Survival
Description: The median survival time, as measured from the start of treatment until death from any cause.
Time Frame: 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Dasatinib Treatment
Number analyzed (Participants) | 15
Months | 27 [1.1 to 47.5]

ADVERSE EVENTS:
Time Frame: From the start of treatment until the participant is taken off study due to disease progression, toxicity, participant withdrawal, or death; median duration of 14 weeks.
Description: Participants were assessed for adverse events with the use of physical exams, laboratory tests, and participant self reporting of adverse events
Arm/Group | Dasatinib Treatment
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 10/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Treatment (N=15)
Neutrophil count decreased (Investigations) | 6
Platelet count decreased (Investigations) | 2
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib Treatment (N=15)
Anemia (Blood and lymphatic system disorders) | 14
Neutrophil count decreased (Investigations) | 7
Platelet Count Decreased (Investigations) | 13
Nausea /vomiting (Gastrointestinal disorders) | 12
Heartburn (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Fatigue (General disorders) | 13
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Headache (Nervous system disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 6
Edema (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes